CLINICAL TRIAL: NCT01826227
Title: Intraoperative Detection of Lesions Using PET (Positron Emission Tomography) Probe During Secondary Cytoreductive Surgery for Recurrent Ovarian, Fallopian Tube and Primary Peritoneal Cancer: A Pilot Study
Brief Title: Intraoperative Detection of Lesions Using PET (Positron Emission Tomography) Probe During Secondary Cytoreductive Surgery for Recurrent Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-017
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2016-12

CONDITIONS: Ovarian Cancer; Fallopian Tube; Primary Peritoneal
Keywords: PET (Positron Emission Tomography); 18F-FDG; Cytoreductive Surgery; 13-017
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Magnetic Resonance Spectroscopy; Cytoreduction Surgical Procedures

ARMS (1):
- Positron Emission Tomography (Experimental): This is a pilot study to determine the ability of intraoperative PET probe to detect and localize recurrent disease. Patients with evidence for a first recurrence of ovarian, fallopian tube or primary peritoneal carcinoma, with evidence of 18F-FDG avid disease on 18F-FDG PET/CT and who are able to undergo secondary CRS are eligible. 20 patients will be studied. All patients will undergo secondary cytoreduction guided by intraoperative PET probe survey. Intraoperative count levels as well as exvivo counts of the resected specimens will be done. Specimens detected with probe only will be labeled so and will be submitted to pathology for histopathologic confirmation.
  Interventions: Procedure: Positron Emission Tomography; Radiation: 18F-Fluoro-2-deoxy-D-lucose; Procedure: Cytoreductive surgery

INTERVENTIONS:
Procedure: Positron Emission Tomography
Radiation: 18F-Fluoro-2-deoxy-D-lucose
Procedure: Cytoreductive surgery

SUMMARY:
The purpose of this study is to see if Positron Emission Tomography (PET) probes make it easier for your surgeon to find cancer and remove it during your surgery. A PET probe is a wandlike device that can detect radioactivity.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of ovarian carcinoma, fallopian tube, or primary peritoneal not to include tumors of low malignant potential (all stage, grade, and histology)
* First recurrence
* Platinum sensitive as defined by disease free interval ≥ 6 months
* Radiological evidence of recurrent disease on preoperative PET/diagnostic CT
* Planned surgical secondary cytoreduction via laparotomy
* >18 years old

Exclusion Criteria:

* Secondary cytoreduction via laparoscopy or robotically assisted laparoscopy
* Tumors of low malignant potential
* Beyond first recurrence
* With the exception of non-melanoma skin cancer, subjects with other invasive malignancies, who had (or have) any evidence of the other cancer present within the last 5 years, are excluded
* Active infection requiring parenteral antibiotics
* For subjects with diabetes mellitus, a blood sugar will be checked preoperatively and must be <200 for participation in the study

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Positron Emission Tomography: This is a pilot study to determine the ability of intraoperative PET probe to detect and localize recurrent disease. Patients with evidence for a first recurrence of ovarian, fallopian tube or primary peritoneal carcinoma, with evidence of 18F-FDG avid disease on 18F-FDG PET/CT and who are able to undergo secondary CRS are eligible. 20 patients will be studied. All patients will undergo secondary cytoreduction guided by intraoperative PET probe survey. Intraoperative count levels as well as exvivo counts of the resected specimens will be done. Specimens detected with probe only will be labeled so and will be submitted to pathology for histopathologic confirmation.
  Positron Emission Tomography
  18F-Fluoro-2-deoxy-D-lucose
  Cytoreductive surgery
Period: Overall Study
Arm/Group | Positron Emission Tomography
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Positron Emission Tomography
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: of detection of lesions with PET probes compared to preoperative FDG18F-FDG PET and standard intraoperative examination. Sensitivity is defined as the percent of lesions that were found with malignant disease divided by the number of lesions with true presence of malignant disease based on the pathology report. A higher sensitivity will indicate a higher number of lesions found with the respective technique thus providing an initial estimate of the incremental benefit of the PET probe as opposed to the other techniques
Time Frame: 2 years
Population: Data not available because the PET probe failed.
Measure: Count of Participants; unit: Participants
Arm/Group | Positron Emission Tomography
Number analyzed (Participants) | 5
Participants | NA — Data not available because the PET probe failed.

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Positron Emission Tomography
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Positron Emission Tomography (N=5)
Supraventricular tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Positron Emission Tomography (N=5)
Anemia (Blood and lymphatic system disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 5
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Blood bilirubin increased (Investigations) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
INR increased (Investigations) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes